CLINICAL TRIAL: NCT01435902
Title: A Randomized, Double-Blind, Double-Dummy, Crossover Comparison of Fluticasone Furoate/Vilanterol 100/25 mcg Once Daily Versus Fluticasone Propionate 250 mcg Twice Daily in Asthmatic Adolescent and Adult Subjects With Exercise-Induced Bronchoconstriction
Brief Title: A Study of a New Asthma Medicine in Asthmatics Whose Asthma Worsens With Exercise
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was cancelled prior to enrolling any subjects
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 106847
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Asthma
Keywords: exercise-induced bronchospasm; Activity/Exercise induced bronchospasm; asthma
MeSH Terms: conditions — Asthma; Asthma, Exercise-Induced; Motor Activity | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone Furoate/Vilanterol (Active Comparator): Fluticasone furoate/vilanterol inhalation powder once daily + Placebo inhalation powder twice daily for 4 weeks
  Interventions: Drug: Fluticasone Furoate/Vilanterol Inhalation Powder
- Fluticasone Propionate (Active Comparator): Fluticasone propionate inhalation powder twice daily + Placebo inhalation powder once daily for 4 weeks
  Interventions: Drug: Fluticasone Propionate Inhalation Powder

INTERVENTIONS:
Drug: Fluticasone Furoate/Vilanterol Inhalation Powder — Fluticasone furoate/Vilanterol inhalation powder inhaled orally once daily for 4 weeks
  Arms: Fluticasone Furoate/Vilanterol
Drug: Fluticasone Propionate Inhalation Powder — Fluticasone propionate inhalation powder inhaled orally twice daily for 4 weeks
  Arms: Fluticasone Propionate

SUMMARY:
The primary objective of this study is to demonstrate that the combination of inhaled fluticasone furoate/vilanterol (100 mcg/25 mcg) once daily provides superior protection throughout the day against bronchoconstriction induced by exercise compared with fluticasone propionate 250 mcg twice daily in adolescent and adult subjects aged 12 to 50 diagnosed with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient male or female 12 to 50 years of age
* Females of child-bearing potential must be willing to use birth control or commit to abstinence during the study
* Diagnosis of persistent asthma for at least 6 months
* Best pre-bronchodilator FEV1 of at least 70%.
* Current use of a low- to moderate-dose inhaled corticosteroid
* Ability to withhold albuterol 6 hours prior to visits.
* Physically able to perform exercise testing on a treadmill when albuterol has been withheld

Exclusion Criteria:

* Intermittent asthma, seasonal asthma, or exercise-induced asthma only
* Symptomatic allergic rhinitis and/or thrush
* Abnormal, clinically significant electrocardigraph
* Respiratory infection within 4 weeks of first visit leading to asthma medication change or could affect subjects's asthma status or participation
* Asthma exacerbation within 12 weeks of first visit
* Respiratory diseases or other concurrent disease that would put subject at risk or confound results interpretation
* Investigational medicines within 30 days of first visit or less than five half-lives of medication in prior study
* Allergy to study drugs or study drug excipients
* Concomitant medications that could interact with study medications or affect the course of asthma
* Tobacco use within last year and/or a 10 pack-years history
* Inability to comply with requirements of the study
* Affiliation with investigator's site (example: family member)

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Maximal percent decrease from baseline in FEV1 following exercise challenge at 12 hours post-dose | At the end of treatment Week 4

SECONDARY OUTCOMES:
Maximal percent decrease from baseline in FEV1 following exercise challenge at 1 hour and 23 hours post-dose | At the end of treatment Week 4
Time required for recovery to within 5% of the pre-exercise baseline FEV1 from the time of the maximal percentage decrease from baseline following the challenge at 1 hour, 12 hours, and 23 hours post-dose | At the end of treatment Week 4
AUC (0-60 minutes) for percentage decrease from baseline in FEV1 after exercise at 1 hour, 12 hours, and 23 hours post-dose | At the end of treatment Week 4
Evaluation of a categorical treatment response using the percentage of subjects who demonstrate a decrease from the pre-exercise baseline in FEV1 of 1) <10%, 2) 10 to <20%, and 3) =/>20%. | At the end of treatment Week 4
Maximal percent decrease from pre-randomized treatment baseline in FEV1 following exercise challenge at 1 hour, 12 hours, and 23 hours post-dose. | At the end of treatment Week 4

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline